CLINICAL TRIAL: NCT01958515
Title: Evaluation of Immunologic Responses in HPV-Associated Oropharyngeal Carcinoma Patients Receiving Chemoradiation Therapy
Brief Title: Immunologic Responses in HPV-Associated Carcinoma for Patients Receiving Chemoradiation
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J13158; IRB00092006 (Other: JHMIRB)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer; HPV (Human Papillomavirus)-Associated Carcinoma; Oropharyngeal
Keywords: Radiation Therapy; Chemotherapy; Chemoradiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chemoradiation with Research Samples: Standard of care chemoradiation therapy will be given as clinically indicated by the treating physicians. 4 research blood and tissue samples will be obtained. One before treatment starts, 2 while treatments are being received and finally one after treatments are completed.
  Interventions: Other: research blood draw and tissue biopsy

INTERVENTIONS:
Other: research blood draw and tissue biopsy — research blood draw and tissue biopsy

SUMMARY:
The primary purpose of this research is to investigate anti-tumor immune responses in patients undergoing chemotherapy and radiation for Head and Neck Cancers.

Hypothesis: Treatment of HPV-associated OPSCC with concurrent chemoradiation results in changes in the tumor microenvironment. We hypothesize that these changes during daily fractionated chemoradiotherapy can lead to detectable changes in HPV-specific tumor immune responses.

Hypothesis: HPV-specific cellular immune responses can still be detected during radiotherapy in the presence or absence of lymphopenia.

* This study will determine whether specific anti-tumor immune responses (Specific Antibodies and Specific T-cells) can be detected in patients undergoing chemoradiation treatment for Head and Neck Cancers.
* This study will evaluate the presence or absence of HPV (human papillomavirus) specific immune responses before, during, and after treatment for Head and Neck Cancers.
* This study will also evaluate whether decreased white blood cell counts may affect development of immune responses in Head and Neck cancer patients undergoing treatment.

Any head and neck cancer patient undergoing concurrent chemoradiotherapy is eligible if: you are older than 18 years of age, capable of providing informed consent, have a life expectancy of greater than 4 months, and have a good performance status.

You are eligible irregardless of your HPV positive or negative status. People with HPV positive (human papillomavirus associated) head and neck cancer may join. People with HPV negative head and neck cancer may also join.

DETAILED DESCRIPTION:
As this is a pilot study seeking to describe the potential impact of chemoradiotherapy on the natural history of any immunologic response in HPV-associated OPSCC, the timing of the venipunctures reflect the goal to sample throughout the course of CTRT (chemoradiation therapy)and will permit some variability based on the number of radiation fractions delivered. It also reflects considerations of time points that lend themselves to both the venipuncture and tumour biopsy based on the toxicity and response profile of the chemoradiation in the HPV-associated OPSCC patient. As such, 10 subjects with HPV-associated OPSCC and 10 subjects with non-HPV associated HNSCC seen by the respective disciplines of otolaryngology-head and neck surgery, radiation oncology, or medical oncology as clinically indicated will be enrolled on this clinical protocol. Importantly, clinical therapeutic recommendations, radiation treatment plans, and therapeutic drugs will not be altered by enrollment in this protocol. Tumors which are directly visible through in office laryngopharyngoscopy and easily accessible (i.e. oropharyngeal tonsil) will be directly biopsied (non-percutaneously) and analyzed as detailed below.

ELIGIBILITY:
Inclusion Criteria:

* patients must have head and neck cancer and be receiving concurrent chemotherapy and radiation
* patients greater than or equal to 18 years of age
* patients must be capable of providing informed consent
* patients must have a life expectancy of greater than 4 months
* patients must have an adequate performance status

Exclusion Criteria:

* Patients must not have had surgery for their head and neck cancer
* Patients must not have a diagnosis of an immunosuppressant disease
* Patients must not have certain uncontrolled concurrent illnesses
* Patients must not a history of autoimmune disease
* Patients must not be pregnant, become pregnant or breast feeding
* Patients must not have a history of certain prior malignancies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 subjects with HPV-associated OPSCC (Oropharyngeal Squamous Cell Carcinoma) and 10 subjects with non-HPV associated HNSCC (Head and Neck Squamous Cell Carcinoma)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Compare Systemic and Local Immunologic Changes During Chemoradiation | Baseline within 1-3 weeks of start of radiation, week 2 between radiation fractions 10-12, week 4 between radiation fractions 20-22, 4-6 weeks after chemoradiation completion
  Primary objective: To evaluate the systemic and local immunologic changes which may occur during a standard treatment course of combined chemoradiation for HPV-associated oropharyngeal squamous cell carcinoma (OPSCC) and non-HPV associated head and neck squamous cell carcinomas (HNSCC).

SECONDARY OUTCOMES:
Relationship of Radiotherapy-Related Lymphopenia and Changes in Cellular Immunity During Chemoradiation | Baseline within 1-3 weeks of start of radiation, week 2 between radiation fractions 10-12, week 4 between radiation fractions 20-22, 4-6 weeks after chemoradiation completion
  Secondary objective: To explore the relationship between radiotherapy-related lymphopenia and changes in cellular immunity during a course of chemoradiation for HPV-associated OPSCC.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Quon, M.D., Principal Investigator — Johns Hopkins SKCCC
Locations (1):
- The Johns Hopkins SKCCC, Baltimore, Maryland, United States